CLINICAL TRIAL: NCT02833805
Title: A Phase II Trial of Non-Myeloablative (NMA) Conditioning and Transplantation of Partially HLA-Mismatched/Haploidentical Related or Matched Unrelated Donor (MUD) Bone Marrow for Newly Diagnosed Patients With Severe Aplastic Anemia
Brief Title: NMA Haplo or MUD BMT for Newly Diagnosed Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1688; IRB00107139 (Other: JHMIRB)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Severe Aplastic Anemia; Aplastic Anemia; Bone Marrow Failure; Immunosuppression
Keywords: immunosuppression; nonmyeloablative; non-myeloablative; allogeneic; tacrolimus; bone marrow; bone marrow transplant; cyclophosphamide; thymoglobulin; ATG; fludarabine
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — thymoglobulin; Antilymphocyte Serum; fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow transplant (Experimental): Non-myeloablative bone marrow transplant with a Thymoglobulin (ATG), fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis.
  Interventions: Drug: Thymoglobulin; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Thymoglobulin — Day -9: 0.5 mg/kg Days -8 and -7: 2 mg/kg daily
  Other Names: Anti-thymocyte globulin; ATG
Drug: Fludarabine — Days -6 through -2: 30 mg/m^2 IV daily
  Other Names: Fludara
Drug: Cyclophosphamide — Days -6 and -5: 14.5 mg/kg IV daily Days 3 and 4: 50 mg/kg IV daily
  Other Names: Cytoxan; Cy; CTX
Radiation: Total body irradiation — Day -1: 200 centigray (cGy) in a single fraction
  Other Names: TBI
Drug: Tacrolimus — Start on Day 5 through Day 365
  Other Names: FK-506; FK506; Prograf
Drug: Mycophenolate mofetil — Days 5 through 35: 15 mg/kg PO three times daily (max 3 g/day)
  Other Names: MMF; CellCept

SUMMARY:
Our primary objective is to determine if it is feasible for previously untreated severe aplastic anemia (SAA) patients to be transplanted using non-myeloablative conditioning and post transplantation cyclophosphamide.

DETAILED DESCRIPTION:
This is a clinical trial of upfront bone marrow transplantation for patients with SAA who do not have a fully human leukocyte antigen (HLA) matched donor. The trial uses a conditioning regimen which has been successful in the refractory and relapsed setting to maximize engraftment and post transplant therapy to minimize graft versus host disease (GVHD). This would be used here in patients who have not yet undergone immunosuppressive therapy for their SAA or are thought to be unlikely to respond to immunosuppressive therapy for SAA.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of inherited or acquired severe aplastic anemia (SAA)
* One of the following available donors:

  1. HLA-haploidentical relative
  2. If recipient is >= 40 years old, may use HLA-matched related donor
  3. For recipients with inherited bone marrow failure syndromes (IBMFS) with clear evidence of same disorder in potential related donors, may use 10/10 matched unrelated donor
* Recipient and/or legal guardian must sign protocol informed consent
* Donor must be willing to donate bone marrow
* Left ventricular ejection fraction (LVEF) >= 40%. For recipients < 13 years old, shortening fraction >= 26% may be used instead.
* Bilirubin < 3 x upper limit of normal (ULN) for age, unless patient has Gilbert's disease
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN for age
* For patients >= 13 years old: estimated creatinine clearance > 50 mL/min using Cockcroft-Gault formula and actual body weight
* For patients >= 1 but < 13 years old: glomerular filtration rate (GFR) estimated by updated Schwartz formula >= 90 mL/min/1.73 m^2. If estimated GFR is < 90 mL/min/1.73 m^2, 24-hour measured creatinine clearance must be > 50 mL/min/1.73 m^2.
* For patients >= 8 years old, diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) > 40%; forced expiratory volume at one second (FEV1) > 50%; forced vital capacity (FVC) > 50%
* For patients < 8 years old or unable to undergo pulmonary function testing: no evidence of dyspnea at rest; no need for supplemental oxygen; oxygen saturation > 92% on room air
* Karnofsky/Lansky status (depending on age) >= 70%
* Females and males of childbearing potential must agree to practice 2 effective methods of contraception at the same time. If unwilling, they must agree to complete abstinence.

Exclusion Criteria:

* Previous administration of immunosuppressive therapy for SAA.
* Fanconi anemia. At minimum, this diagnosis must be excluded by diepoxybutane (DEB) or equivalent testing on peripheral blood or marrow in patients < 30 years old.
* Clonal cytogenetic abnormalities consistent with pre-myelodysplastic syndrome (pre-MDS) or MDS on bone marrow examination
* Presence of anti-donor antibodies
* Prior allogeneic stem cell transplant
* Prior solid organ transplant
* Uncontrolled bacterial, viral, or fungal infection
* HIV seropositivity
* Active hepatitis B or C infection determined by serology and/or nucleic acid testing (NAT)
* Pregnancy or active breastfeeding
* Prior malignancies except: resected basal carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent > 5 years previously. Other prior cancers will not be allowed unless approved by the PI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy E DeZern, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeZern AE, Zahurak M, Symons HJ, Cooke KR, Huff CA, Jain T, Swinnen LJ, Imus PH, Wagner-Johnston ND, Ambinder RF, Levis M, Luznik L, Bolanos-Meade J, Fuchs EJ, Jones RJ, Brodsky RA. Alternative donor BMT with posttransplant cyclophosphamide as initial therapy for acquired severe aplastic anemia. Blood. 2023 Jun 22;141(25):3031-3038. doi: 10.1182/blood.2023020435. PMID 37084383
- [Derived] DeZern AE, Zahurak ML, Symons HJ, Cooke KR, Rosner GL, Gladstone DE, Huff CA, Swinnen LJ, Imus P, Borrello I, Wagner-Johnston N, Ambinder RF, Luznik L, Bolanos-Meade J, Fuchs EJ, Jones RJ, Brodsky RA. Haploidentical BMT for severe aplastic anemia with intensive GVHD prophylaxis including posttransplant cyclophosphamide. Blood Adv. 2020 Apr 28;4(8):1770-1779. doi: 10.1182/bloodadvances.2020001729. PMID 32343796

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Transplant: Non-myeloablative bone marrow transplant with a Thymoglobulin (ATG), fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as graft-versus-host disease (GVHD) prophylaxis.
  Thymoglobulin: Day -9: 0.5 mg/kg Days -8 and -7: 2 mg/kg daily
  Fludarabine: Days -6 through -2: 30 mg/m^2 IV daily
  Cyclophosphamide: Days -6 and -5: 14.5 mg/kg IV daily Days 3 and 4: 50 mg/kg IV daily
  Total body irradiation: Day -1: 200 centigray (cGy) in a single fraction
  Tacrolimus: Start on Day 5 through Day 365
  Mycophenolate mofetil: Days 5 through 35: 15 mg/kg PO three times daily (max 3 g/day)
Period: Overall Study
Arm/Group | Bone Marrow Transplant
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [3 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4
  Caucasian | 14
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival and Engraftment at One Year
Description: Number of enrolled participants who receive BMT, achieve engraftment, and are alive at one year post bone marrow transplant (BMT).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 19

2. Secondary Outcome: Overall Survival at One Year
Description: Number of participants alive at one year after BMT.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 19

3. Secondary Outcome: Probability of Neutrophil Recovery as Assessed by the Number of Participants Who Have Recovered Neutrophil Counts
Description: Probability of neutrophil recovery will be assessed by the number of participants who have recovered neutrophil counts at 1 year (>500 ANC).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 21

4. Secondary Outcome: Probability of Platelet Recovery as Assessed by Number of Participants Who Have Recovered Platelet Counts
Description: Probability of platelet recovery will be assessed by the number of participants who have recovered platelet counts at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 20

5. Secondary Outcome: Number of Participants Who Experience Primary Graft Failure
Description: Number of participants who experience primary graft failure by one year after BMT.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 21

6. Secondary Outcome: Number of Participants Who Experience Secondary Graft Failure
Description: Number of participants who experience secondary graft failure by one year after BMT.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 19

7. Secondary Outcome: Number of Participants Who Experience Grades II-IV Acute GVHD
Description: Number of participants who experience grade II, III, or IV acute GVHD by Day 100.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 4

8. Secondary Outcome: Number of Participants Who Experience Grades III-IV Acute GVHD
Description: Number of participants who experience grade III or IV acute GVHD by Day 100.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 2

9. Secondary Outcome: Number of Participants Who Experience Chronic GVHD
Description: Number of participants who experience chronic GVHD by two years after BMT.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 1

10. Secondary Outcome: Number of Participants With Full Donor Chimerism
Description: Number of participants with full donor chimerism at Day 60.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 21

11. Secondary Outcome: GVHD-free Relapse-free Survival (GRFS)
Description: Number of participants alive, without relapse, and without GVHD at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 19

12. Secondary Outcome: Transplant-related Mortality
Description: Number of participants deceased for reasons related to BMT at 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 21
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected from time of consent up to one year.
Arm/Group | Bone Marrow Transplant
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bone Marrow Transplant (N=21)
Gram negative rods Bacteremia (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02833805/Prot_SAP_000.pdf